CLINICAL TRIAL: NCT05529225
Title: Evaluating the Usability, Efficacy and Commercial Utility of a Digital Platform to Deliver Comprehensive Treatment for Opioid Use Disorder
Brief Title: Evaluating the Efficacy of a Digital Platform to Deliver Comprehensive Treatment for Opioid Use Disorder
Acronym: BEaTS
Status: Completed | Type: Observational
Sponsor: Boulder Care (Industry)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: 1R44DA050354-02 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2022-09-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; Telehealth; Retention in Care
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Boulder Care: People seeking buprenorphine for opioid use disorder via telehealth.
- OHSU: People seeking buprenorphine for opioid use disorder via treatment as usual.

SUMMARY:
Buprenorphine Evaluation and Telehealth Study (BEaTS)

Comparison of retention in care between telehealth-based care and treatment as usual.

DETAILED DESCRIPTION:
Evaluating the Usability, Efficacy and Commercial Utility of a Digital Platform to Deliver Comprehensive Treatment for Opioid Use Disorder

Phase I, Aim I: Completed (R44 DA050354). Advance Boulder Care's mobile platform development and obtain usability feedback from individuals with prior OUD treatment. Aim 1 was successfully completed during Phase I, meeting milestones for improving product usability and satisfaction while reducing treatment barriers.

Phase II, Aim 2: Compare study participants who enroll in Boulder Care (n = 100) to participants who enroll in treatment as usual (i.e., office-based buprenorphine) (n = 100) and assess buprenorphine retention at 48 weeks (primary outcome) and monitor a) transition from referral to treatment, b) care continuity, c) engagement in care, and d) satisfaction with care (secondary outcomes).

Phase II, Aim 3: Compare study participants who enroll in Boulder Care (n = 100) to participants who enroll in treatment as usual (i.e., office-based buprenorphine) (n = 100) and assess at baseline, 4, 12, 24, 36, and 48 weeks post treatment initiation opioid use (primary outcome) and monitor employment, housing stability, and criminal justice involvement (secondary outcomes).

Phase II Approach.

The COVID-19 pandemic has altered treatment and research for OUD. Phase II of the Small Business Innovation Research (SBIR) award "Evaluating the usability, feasibility and commercial utility of a digital platform to deliver comprehensive treatment for opioid use disorder" (R44 DA050354) takes advantage of further development of the Boulder Care platform and expands the testing of our digitally-delivered treatment.

To assure the quality and success of the Phase II award, a partnership with experienced National Institute on Drug Abuse (NIDA) investigators under the leadership of Todd Korthuis, MD, MPH, strengthens the application. The application is modified to take advantage of Dr. Korthuis' and his team's experience and access to the Oregon Health & Science University (OHSU) Harm Reduction and Bridges to Recovery clinic (HRBR - pronounced "harbor") and buprenorphine prescribing at OHSU primary care clinics. The HRBR clinic offers low-barrier buprenorphine initiation and stabilization, linking patients to community providers for ongoing care. The clinic can provide referrals to facilitate recruitment to Boulder Care services and participation in the Phase II study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with a diagnosis of OUD
* Within 45 days of seeking buprenorphine prescription
* Have a working smartphone
* Speaks and understands English

Exclusion Criteria:

* Untreated mental or medical health conditions that, in the opinion of the patient, would preclude study participation
* History of allergic reaction to buprenorphine
* Impending incarceration
* Plans to move out of Oregon in next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People seeking buprenorphine treatment for opioid use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Retention in treatment | 48 weeks
  The primary Goal of the Phase II project is to compare participant retention in buprenorphine treatment for opioid use disorder (OUD) at 48 weeks for participants enrolled in Boulder Care (n=l00) to participants enrolled in treatment-as-usual (TAU) from OHSU (Oregon Health & Science University) clinics (n=100).
  Retention in treatment will be assessed through the Electronic Medical Record for each patient and whether there is an active buprenorphine prescription for the patient at 48 weeks of care. Because of the protocols for each clinic, such a prescription will indicate that treatment is active for a given participant.
  This is the most direct way to assess ongoing buprenorphine treatment as Oregon law prohibits use of its Prescription Drug Monitoring Program for research.

SECONDARY OUTCOMES:
Participant satisfaction | 48 weeks
  Participant satisfaction with telehealth comparing Boulder Care's fully digital integrated platform to OHSU's TAU approach which uses in-person treatment as well as ad-hoc telehealth due to the COVID-19 pandemic.
  Assessment at baseline and weeks 4, 12, 24, 36 and 48 after enrollment in the study.
  Patient satisfaction with treatment is assessed via a single-item: "How satisfied are you with your buprenorphine treatment?" with 5-point Likert scale (very dissatisfied, dissatisfied, neither satisfied nor dissatisfied, satisfied, very satisfied) adapted from treatment satisfaction measures used in the National Drug Abuse Treatment Clinical Trials Network studies.
Changes in cravings, health perception, and health care utilization | 48 weeks
  Changes in cravings, health perception, and health care utilization.
  Assessment at baseline and weeks 4, 12, 24, 36 and 48 after enrollment in the study.
  Degree of craving will be assessed with the 17-item Brief Addiction Monitor (BAM) and the 4-item Treatment Effectiveness Assessment (TEA). Health perception will be assessed with the CDC's health-related quality of life (HRQoL) instrument. Health care utilization will be assessed from the medical record and patient report.
Changes in risk factors for substance use and for protective factors that support recovery | 48 weeks
  Changes in risk factors for substance use and for protective factors that support recovery.
  Assessment at baseline and weeks 4, 12, 24, 36 and 48 after enrollment in the study.
  The 17-item Brief Addiction Monitor (BAM) and the 4-item Treatment Effectiveness Assessment (TEA) will be used to evaluate these risk and protective factors.
Changes in demographics i.e., employment, education, housing, etc | 48 weeks
  Changes in demographics i.e., employment, education, housing, etc.
  Assessment at baseline and weeks 4, 12, 24, 36 and 48 after enrollment in the study.
  We assess functional outcome measures using the 17-item Brief Addiction Monitor (BAM), and the 4-item Treatment Effectiveness Assessment (TEA). These instruments incorporate patient-centered functional measures of recovery such as relationships, employment, spiritual comfort, and achievement of self-identified treatment goals in addition to assessments of drug use.

OTHER OUTCOMES:
Evaluation of opioid use | 48 weeks
  A second goal is to compare study participants from Boulder care to OHSU TAU participants for opioid use at baseline, 4, 12, 24, 36, and 48 weeks post study enrollment.
  Self-reported use of any opioids (heroin, fentanyl, other non-prescribed opioids), will be derived from Addiction Severity Index-Lite (ASI-Lite) drug use questions and adapted to assess the number of days of use in the past 28 days. The primary outcome measure is dichotomized as ≥1 day of use versus no days of use at 48 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Strong, Principal Investigator — Boulder Care
Locations (2):
- United States (2):
  - Boulder Care, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No